CLINICAL TRIAL: NCT06165159
Title: Influence du Type de Traitement du diabète de Type 1 (DT1) Sur la Charge Mentale Des Adolescents Avec un DT1 et Des Parents Ayant un Enfant Avec DT1.
Brief Title: Influence of Type 1 Diabetes (T1DM) Treatment Type on Mental Workload
Acronym: CHAM&DIAB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0257
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes; Treatment
Keywords: Type 1 diabetes; Children; Adolescents; Parents; Pump; Multiple injections; Closed loop; Burden of treatment; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: children and adolescents with type 1 diabetes and their parents — "Children over the age of 8 with type 1 diabetes diagnosed more than 6 months ago in France, followed in one of the hospitals that are members of the Aide aux Jeunes Diabétiques (AJD) association.
  Parents or people involved in the day-to-day life of children with type 1 diabetes diagnosed at least 6 months ago, whose child is being followed in France in one of the hospitals affiliated to the AJD association."

SUMMARY:
Influence of the type of treatment for type 1 diabetes (pump versus multiple injections versus closed loop) on the treatment burden of children and adolescents and their parents.

DETAILED DESCRIPTION:
"The guidelines for the treatment of children and adolescents with type 1 diabetes emphasise an individualised approach to the child and provide target values (time in range, glycaemia and coefficient of variation). These recommendations aim to prevent long-term complications. It is rarely possible to achieve and maintain this level of control over the long term. Achieving these recommendations requires a great deal of investment from children and their families, which can significantly increase their psychological workload and reduce their quality of life.

The main aim of this study was to assess burden of treatment according to the treatment type (pump versus multiple injections versus closed loop) on a large scale."

ELIGIBILITY:
Inclusion Criteria:

* Children over the age of 8 whose type 1 diabetes has been diagnosed for at least 6 months
* Parents or people involved in the day-to-day life of children with type 1 diabetes who have been diagnosed for at least 6 months

Exclusion Criteria:

* Parents not involved in managing their child's type 1 diabetes (child in care)
* Have already completed the questionnaire (one questionnaire completed per child and their parents or family caregivers)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the national network of the Association d'Aide aux Jeunes Diabetiques (AJD). The AJD federates local patient associations, which are regularly asked to distribute questionnaires to their members.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome corresponds to the score obtained after completing the study questionnaire. The questionnaire is completed at the participation agreement. | 1 day
  The primary outcome is the treatment burden according to the treatment modality (semi-closed loop versus insulin pump versus multi-injection) assessed using a specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle LABARRE, Principal Investigator — Angers University Hospital
Locations (1):
- Emmanuelle LABARRE, Angers, France